CLINICAL TRIAL: NCT05651204
Title: Electrophysiological Biomarkers of GABA Metabolism in Children With SCN1A+ Dravet Syndrome
Brief Title: GABA Biomarkers in Dravet Syndrome
Status: Recruiting | Type: Observational
Sponsor: Cook Children's Health Care System (Other)
Collaborators: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-051
Record Dates: First submitted 2022-10-07; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dravet
  Interventions: Diagnostic Test: GABA Blood Level
- Age-Matched Control
  Interventions: Diagnostic Test: GABA Blood Level

INTERVENTIONS:
Diagnostic Test: GABA Blood Level — Blood specimens will be collected by a registered phlebotomist according to hospital's specimen collection procedures.

SUMMARY:
This study will non-invasively obtain levels of GABA in the brain of children with SCN1A+DS and neurodeveloping children through evoked and induced cortical responses, correlate them with the BOLD responses, and with the levels of GABA in their blood.

DETAILED DESCRIPTION:
Epileptic seizures may result from too much excitation or too little inhibition in the area in which abnormal discharges start. Excitation and inhibition of neurons are mediated by g-aminobutyric acid (GABA) neurotransmitter among others. Several lines of evidence indicate an abnormal pathophysiological mechanism of GABA in children with Dravet Syndrome (DS). Other studies show that measures of the beta and gamma brain activity with non-invasive electrophysiological techniques correlate with the levels of GABA in the human brain. Here, we propose to assess these measures in children with SCN1A+DS and neurodeveloping healthy controls aiming to develop noninvasive biomarkers for the monitoring of the levels of GABA in their brain. Such a biomarker would be useful for understanding the pathophysiological GABA mechanism in children with DS and potentially guide the development of future GABAergic modulation treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Authorized representative (parent/caregiver) must be willing and able to give informed consent for the participant's participation in the study. Participants capable of providing informed assent must be willing to provide their assent.
2. Participant and their parent/caregiver are willing and able (in the PI's opinion) to comply with all study requirements.
3. Participant is male or female aged between 0 months and 18 years of age, inclusive, at the time of consent.
4. Participant has a confirmed pathogenic or likely pathogenic SCN1A mutation, as demonstrated by genetic testing.
5. Participant had normal development prior to onset of first seizure as defined by the Centers for Disease Control and Prevention (CDC 2019).
6. Participant had an onset of seizures, defined as first focal clonic/hemiclonic, generalized/focal, generalized tonic-clonic/clonic, atonic, prolonged seizure, or status epilepticus between age 3 and 5 months, inclusive.
7. Participant should have an evaluation by a pediatric neurologist with a diagnosis of DS.

Exclusion Criteria:

1. Participant has a copy number variant of SCN1A, including SCN1A microdeletion, affecting other genes.
2. Participant has an SCN1A mutation present on both alleles.
3. Participant has a known pathogenic or clinically suspected mutation in a seizure-associated gene besides SCN1A.
4. Participant has a confirmed mutation in a gene besides SCN1A, that is known to increase the severity of the seizure phenotype.
5. Participant has a known gain-of-function mutation, as defined by functional studies, including p.Thr226Met.
6. Participant has a history of notable developmental deficit that was evident prior to seizure onset, by physician report.
7. Participant has a known central nervous system structural abnormality as found on magnetic resonance imaging or computed tomography scan of brain which, in the opinion of the Principal Investigator (PI), is not consistent with the clinical phenotype of DS. Note: Prior scans may be used, and no new scan is required to confirm normal imaging.
8. Metal implants.
9. Baclofen pump.
10. Inability or unwillingness of patient or parent/legally authorized representative to give written informed consent (and/or assent as appropriate).

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will recruit 18 children with a diagnosis of SCN1A+DS and 18 aged-matched neurotypical children (all aged 0-18 years old).
  Participants will be divided into three different age groups:
  * 0-7 years old (n=12; 6 children with a diagnosis of SCN1A+ DS and 6 age-matched neurotypical children).
  * >7-12 years old (n=12; 6 children with a diagnosis of SCN1A+ DS and 6 age-matched neurotypical children).
  * >12-18 years old (n=12; 6 children with a diagnosis of SCN1A+ DS and 6 age-matched neurotypical children).
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-09-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
GABA Blood Level | Up to 30 minutes
  GABA levels evaluated by clinical blood draw.

SECONDARY OUTCOMES:
BOLD (Blood oxygenation level dependent) MRI | Up to 1.5 hours
  For the task-fMRI scans, we will present to the participant child-friendly cartoon images and videos in order to localize the visually-induced BOLD response in their primary visual cortex. We will also deliver compressed air-puffs using a pneumatic stimulator and brush their fingers with a toothbrush in order to localize the somatosensory-induced BOLD response in their primary somatosensory cortex. Lastly, we will deliver to the participant beep sounds through an MRI-compatible headset in order to localize the auditory-induced BOLD response in their primary auditory cortex.
MEG | Up to 3 hours
  We will use the MEG to measure evoked fields and potentials elicited by somatosensory, auditory, and visual stimuli.
HD-EEG | Up to 90 minutes
  We will use HD-EEG to measure evoked fields and potentials elicited by somatosensory, auditory, and visual stimuli.
TMS | Up to 2 Hours
  TMS is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain in order to map the motor cortex. An electromagnetic coil is placed against the scalp near the forehead. The electromagnet non-invasively delivers a magnetic pulse that stimulates nerve cells in the region of your brain involved in motor control.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Papadelis, PhD, Principal Investigator — Cook Children's Health Care System
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No